CLINICAL TRIAL: NCT07334873
Title: Evaluation of the Efficacy of Inhaled Nitric Oxide Therapy in Patients With Moderate to Severe Acute Respiratory Distress Syndrome: A Multicenter, Prospective, Randomized Controlled Clinical Trial (ENARCT-ARDS)
Brief Title: Effect of Inhaled Nitric Oxide Therapy in Adults With Moderate-to-Severe Acute Respiratory Distress Syndrome
Acronym: ENARCT-ARDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NFEC-2025-708
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: ARDS (Moderate or Severe)
Keywords: Inhaled Nitric Oxide Therapy; ARDS
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care for ARDS+Inhaled Nitric Oxide (Experimental)
  Interventions: Procedure: Inhaled Nitric Oxide Therapy

INTERVENTIONS:
Procedure: Inhaled Nitric Oxide Therapy — Patients randomized to the intervention group will receive inhaled nitric oxide (iNO) delivered via the portable INOwill N200 system in addition to standard ARDS care. iNO administration will commence immediately upon enrollment, with its concentration set and titrated in accordance with established clinical practice guidelines.

SUMMARY:
The goal of this clinical trial is to evaluate whether inhaled nitric oxide (iNO), added to standard care, can reduce mortality in adults with moderate-to-severe Acute Respiratory Distress Syndrome (ARDS). The main questions it aims to answer are:

Does iNO therapy reduce 28-day all-cause mortality compared to standard care alone? Does iNO therapy increase the number of ventilator-free days through day 28? If there is a comparison group: Researchers will compare the group receiving iNO plus standard care with the group receiving placebo plus standard care to see if iNO improves survival and other clinical outcomes.

Participants will:

Be randomly assigned to receive either iNO or a placebo through the ventilator.

Receive all other standard treatments for ARDS as per current guidelines. Be closely monitored for 28 days to track survival, time on the ventilator, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients diagnosed with moderate-to-severe ARDS according to the 2023 Global (or international) criteria.

Exclusion Criteria:

* Known allergy to iNO.
* Congenital methemoglobinemia.
* End-stage chronic lung disease (e.g., lung cancer, prior pneumonectomy/lung transplant).
* Shock (norepinephrine >0.5 μg/kg/min or equivalent for >6 hours) at treatment initiation.
* Pulmonary hypertension (PASP >45 mmHg by echo or mPAP ≥25 mmHg by catheterization).
* Serum creatinine >2.5 mg/dL (221 μmol/L).
* Major bleeding (e.g., intracranial, pulmonary) or platelet count <20×10⁹/L.
* Expected ICU/mechanical ventilation <24 hours.
* Pre-enrollment ECMO therapy.
* Any investigator-assessed unsuitability for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | within 28 days after randomization
  The primary outcome was 28-day all-cause mortality, defined as death from any cause occurring within 28 days following randomization. All patients must be followed up through day 28, regardless of hospital discharge status.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided